CLINICAL TRIAL: NCT00546286
Title: A 12 Week, Open-Label, Study to Evaluate the Effectiveness of Dorzolamide-Timolol as First Line Therapy to Reduce Intraocular Pressure in Patients With Untreated Open Angle Glaucoma (OAG) or Ocular Hypertension (OH)
Brief Title: A Study to Evaluate the Effectiveness of Cosopt® as First Line Therapy (MK-0507A-153)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0507A-153; MK0507A-153; 2007_027
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — dorzolamide-timolol combination; Prostaglandins

ARMS (2):
- 1 (Experimental): dorzolamide HCl/timolol maleate
  Interventions: Drug: dorzolamide hydrochloride (+) timolol maleate
- 2 (Experimental): dorzolamide hydrochloride/timolol maleate + prostaglandin
  Interventions: Drug: Comparator: dorzolamide HCl/timolol maleate + prostaglandin

INTERVENTIONS:
Drug: dorzolamide hydrochloride (+) timolol maleate — Combination treatment of dorzolamide HCl (2%)/ timolol maleate (0.5%) BID for six weeks in patients with open-angle glaucoma or ocular hypertension.
  For patients who achieve target IOP at 6 weeks, dorzolamide/timolol is continued for another 6 weeks.
  Other Names: Cosopt
  Arms: 1
Drug: Comparator: dorzolamide HCl/timolol maleate + prostaglandin — Combination treatment of dorzolamide HCl (2%)/timolol maleate(0.5%) BID for six weeks in patients with open-angle glaucoma or ocular hypertension.
  For patients not achieving target IOP at 6 weeks, a prostaglandin is added for another 6 weeks.
  Other Names: Cosopt
  Arms: 2

SUMMARY:
Evaluate the effectiveness of dorzolamide-timolol (Cosopt®) as first line therapy in reducing intraocular pressure in patients with untreated Open angle glaucoma (OAG) or Ocular hypertension (OH).

ELIGIBILITY:
Inclusion Criteria:

* Patient has been recently diagnosed and is presently untreated for Open-Angle Glaucoma Or Ocular Hypertension With An iop of at least 27 mmhg in at least one eye (patient's worse eye)
* Patient Already Diagnosed With Open-Angle Glaucoma Or Ocular Hypertension And Untreated For At Least 30 Days Are Eligible For The Study If They Have An Iop Of 27 Mmhg Or More In At Least One Eye

Exclusion Criteria:

* A History Of Any Illness That, In The Opinion Of The Investigator, Might Confound The Results Of The Study Or Pose Additional Risk By Administering Dorzolamide-Timolol (Cosopt®) Or Prostaglandins
* The Presence Of Any Fundus Pathology Likely To Change During The Study Or To Influence Iop (Background Of Diabetic Retinopathy Is Permitted)
* Any Contraindication To The Use Of Cosopt® Including: - Bronchospasm, Including Bronchial Asthma Or A History Of Bronchial Asthma Or Chronic Obstructive Pulmonary Disease. - Sinus Bradycardia, Second Or Third Degree Av Block, Cardiac Failure (Grade Iii And Iv), Cardiogenic Shock
* Patient On Oral Carbonic Anhydrase Inhibitor, Concomitant Systemic Or Dermatological Medication Known To Affect The Iop, E.G. Clonidine, Corticosteroids, Oral Beta-Blocking Agents
* Pregnant Woman Or A Woman Of Childbearing Potential Who Is Sexually Active And Not Using An Acceptable Method Of Contraception (For Ex: Oral Contraceptive, Diaphragm, Contraceptive Sponge, Intra-Uterine Device, Long-Acting Contraceptive Injections, Double-Barrier Methods) Beginning At Least 7 Days Prior To Treatment And Continuing At Least 14 Days After The Last Visit Or The Discontinuation Visit. (Women Who Are Postmenopausal Or Have Received A Hysterectomy Or Have Undergone Tubal Ligature Are Considered As Not Having Childbearing Potential.)
* Severe Renal Impairment (Serum Creatinine > 150 umol/L Or Creatinine Clearance < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-05-31 (Actual); Primary Completion 2007-08-23 (Actual); Study Completion 2007-08-23 (Actual)

PRIMARY OUTCOMES:
Reduction in IOP 4 mmHg (or >= 20%) over a period of 6 or 12 weeks. | 6 to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Crichton AC, Harasymowycz P, Hutnik CM, Behki R, Boucher S, Ibrahim F, Rifkind AW, Solomon L, Liao C, Bastien NR, Sampalis JS. Effectiveness of dorzolamide-timolol (COSOPT) in patients who were treatment naive for open-angle glaucoma or ocular hypertension: the COSOPT first-line study. J Ocul Pharmacol Ther. 2010 Oct;26(5):503-11. doi: 10.1089/jop.2010.0032. PMID 20874498
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html